CLINICAL TRIAL: NCT02766946
Title: Ultrasound Observation of Diaphragmatic Atrophy Related to Mechanical Ventilation A Prospective Monocentric Study in Intensive Care Unit
Brief Title: Diaphragmatic Atrophy Related to Mechanical Ventilation
Acronym: ECHODIAPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SJSL12013
Record Dates: First submitted 2016-04-29; First posted 2016-05-10 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Septic Shock; Acute Respiratory Distress
Keywords: Mechanical Ventilation
MeSH Terms: conditions — Shock, Septic; Acute Lung Injury | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mechanical Ventilation (Experimental): Evolution over time of Diaphragmatic and Pectoralis muscle atrophy under Mechanical Ventilation
  Interventions :
  * Ultrasound of the right diaphragm
  * Ultrasound of the pectoral muscle
  * Neuromyopathy score
  * Respiratory performances
  Interventions: Device: Ultrasound; Other: Neuromyopathy score; Other: Respiratory performances
- Non-invasive Ventilation (Active Comparator): Evolution over time of Diaphragmatic and Pectoralis muscle atrophy under Non-invasive Ventilation
  Interventions :
  * Ultrasound of the right diaphragm
  * Ultrasound of the pectoral muscle
  * Neuromyopathy score
  * Respiratory performances
  Interventions: Device: Ultrasound; Other: Neuromyopathy score; Other: Respiratory performances
- Spontaneous Ventilation (Active Comparator): Evolution over time of Diaphragmatic and Pectoralis muscle atrophy under Spontaneous Ventilation
  Interventions :
  * Ultrasound of the right diaphragm
  * Ultrasound of the pectoral muscle
  * Neuromyopathy score
  * Respiratory performances
  Interventions: Device: Ultrasound; Other: Neuromyopathy score; Other: Respiratory performances

INTERVENTIONS:
Device: Ultrasound — An ultrasound of the right diaphragm will be performed on day 1, day 3, day 5 and day 10
Device: Ultrasound — An ultrasound of the pectoral muscle will be performed on day 1, day 3, day 5 and day 10
Other: Neuromyopathy score — A neuromyopathy score will be assessed on the extubation day
Other: Respiratory performances — An assessment of the respiratory performances will be done on the extubation day, including higher expiratory pressure, higher inspiratory pressure, and occlusion pressure

SUMMARY:
Ventilatory support during critical phase result in inactivity of respiratory muscles especially diaphragm muscle. These inactivity also result in change of contractile capability and quick muscular atrophy.

The aim of the study is to visualize the evolution of diaphragm thickness by echography during Mechanical Ventilation for patients with septic shock or acute respiratory distress syndrome and to compare with the evolution for patients under non-invasive ventilation and those with spontaneous ventilation. Measurements will be performed at day 1, day 5 and day 10 (if patient still under a mode of ventilation or in the unit).

The evolution of diaphragm thickness will also be compared to pectoralis muscle atrophy, which is not involved in ventilation, in order to assess respective effect of ventilatory inactivity and undernutrition linked to intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Group 1 : under Mechanical Ventilation (time of Mechanical Ventilation for at least 5 days)
* Group 2 : under Non-invasive Ventilation
* Group 3 : Spontaneous Ventilation
* Non opposition of patient (Groups 2 and 3) or non-opposition of patient family member (Group 1)

Exclusion Criteria:

* Known diaphragmatic paralysis
* Neurologic pathology with motor deficit
* Pregnancy or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2013-06-24 (Actual); Primary Completion 2015-12-17 (Actual); Study Completion 2015-12-22 (Actual)

PRIMARY OUTCOMES:
Change from day 1 diaphragm thickness at day 3 and day 5 | 1 day, 3 days and 5 days after introduction of Mechanical Ventilation
  Diaphragm thickness measured by ultrasound

SECONDARY OUTCOMES:
Diaphragm thickness measured by ultrasound | 10 days after introduction of Mechanical Ventilation
Type of ventilatory support | 10 days after start of ventilatory support
  Define which type of ventilatory support is used (mechanical ventilation, non-invasive ventilation, or spontaneous ventilation)
Ventilatory mode | 10 days after start of ventilatory support
  Ventilatory mode (controlled ventilation, pressure support ventilation)
Pectoralis muscle thickness measured by ultrasound | 10 days after start of ventilatory support
  To compare the importance of this atrophy to those of diaphragmatic muscle
Diaphragmatic strength | intraoperative
  Relation between diaphragmatic atrophy and decrease of diaphragmatic strength
Early or late extubation failure rate (extubation performed before or after 48 hours) | The last day of hospitalisation
  Relation between diaphragmatic atrophy importance and premature (<48h) or late extubation failure
MRC score (Medical Research Council) | intraoperative
  Relation between diaphragmatic atrophy and decrease of diaphragmatic strength
Length of ventilation in hours | 10 days after start of ventilatory support
Drug administration | 10 days after start of ventilatory support
  Presence of drug administration such as curare, corticoid or sedative. If yes : number of days with treatment
Total positive end expiratory pressure | 10 days after start of ventilatory support
External positive end expiratory pressure | 10 days after start of ventilatory support
Respiratory rate | 10 days after start of ventilatory support
Highest inspiratory pressure level | 10 days after start of ventilatory support
Highest expiratory pressure level | 10 days after start of ventilatory support
Volume of exhaled air | 10 days after start of ventilatory support